CLINICAL TRIAL: NCT02433236
Title: A Phase 2, Multi-Centre, Open Label Extension Study of Fostamatinib in the Treatment of IgA Nephropathy for Patients Who Participated in Study C-935788-050
Brief Title: Open Label Study of Fostamatinib in the Treatment of IgA Nephropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment of first subject
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-935788-051
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: IGA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fostamatinib Disodium tablet 100 mg (Experimental): Fostamatinib Disodium tablet 100 milligram (mg) by mouth twice a day for 15 months
  Interventions: Drug: Fostamatinib Disodium tablet 100 mg
- Fostamatinib Disodium tablet 150 mg (Experimental): Fostamatinib Disodium tablet 150 milligram (mg) by mouth twice a day for 15 months
  Interventions: Drug: Fostamatinib Disodium tablet 150 mg

INTERVENTIONS:
Drug: Fostamatinib Disodium tablet 100 mg
  Other Names: Fostamatinib; R788
  Arms: Fostamatinib Disodium tablet 100 mg
Drug: Fostamatinib Disodium tablet 150 mg
  Other Names: Fostamatinib; R788
  Arms: Fostamatinib Disodium tablet 150 mg

SUMMARY:
Phase 2, multi-center, open label extension study to evaluate 2 dose regimens of fostamatinib in approximately 25 subjects. The study will consist of 11 visits over 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study C-938788-050, including having received a post-treatment renal biopsy, and having had a clinically meaningful response (i.e. decreased proteinuria or improved renal histology)
* Able and willing to give written informed consent

Exclusion Criteria:

* Unresolved Grade 2 or greater toxicity in Study C-935788-050

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with mean change of Proteinuria as measured by spot urine protein/creatinine ratio (sPCR) | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Rigel Pharmaceuticals, Inc., Study Director — Rigel Pharmaceuticals,Inc.